CLINICAL TRIAL: NCT04763434
Title: Dexamethasone and Dexmedetomidine as Adjuvants to Ropivacaine in Ultrasound-guided Multilevel Thoracic Paravertebral Block for Lobectomy: A Prospective, Randomized, Triple-blind Study
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Gansu Provincial Hospital (Other)
Responsible Party: Principal Investigator, dong zhang, dong zhang, Gansu Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GanSu provincial hospital
Record Dates: First submitted 2021-02-17; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Dexamethasone; Dexmedetomidine; Ropivacaine; Lobectomy
MeSH Terms: interventions — Dexamethasone; Dexmedetomidine; Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- RS group (Active Comparator): 20 ml mixture of 37.5 mg ropivacaine with 5 mg dexamethasone
  Interventions: Drug: dexamethasone; dexmedetomidine; ropivacaine
- RM group (Active Comparator): 20 ml mixture of 37.5 mg ropivacaine with 1 µg/kg dexmedetomidine
  Interventions: Drug: dexamethasone; dexmedetomidine; ropivacaine
- RSM group (Experimental): 20 ml mixture of 37.5 mg ropivacaine with 1 µg/kg dexmedetomidine and 5 mg dexamethasone (RSM group)
  Interventions: Drug: dexamethasone; dexmedetomidine; ropivacaine

INTERVENTIONS:
Drug: dexamethasone; dexmedetomidine; ropivacaine — Ultrasound-guided multilevelTPVB is performed at the end of lobectomy

SUMMARY:
The hypothesis is whether perineural dexamethasone and dexmedetomidine prolonged the duration of analgesia as compared with either perineural dexamethasone or perineural dexmedetomidine after TPVB.

DETAILED DESCRIPTION:
Design: A prospective, randomized, controlled study Setting: Single-center university hospital. Participants: The study included 90 patients undergoing lobectomy under general anesthesia.

Interventions: The patients were allocated randomly into the following 3 groups: 20 ml mixture of 37.5 mg ropivacaine with 5 mg dexamethasone (RS group) or 1 µg/kg dexmedetomidine (RM group), or with 1 µg/kg dexmedetomidine and 5 mg dexamethasone (RSM group). Ultrasound-guided TPVB was performed at 4 points-T4-5, T5-6, T6-7, and T7-8 of the surgical side; 5 mL of solution were injected at each point. Postoperatively, the PCIA was used as part of multimodal analgesia, and all patients recieve .

ELIGIBILITY:
Inclusion Criteria:

ASA physical status I-II grade Undergoing elective lobectomy under general anesthesia. Participants aged from 16-65 years old.

Exclusion Criteria:

Refusal for TPVB Inability to obtain informed consent Coagulation disorders, neuropathy, or body mass index greater than 40 kg/m2 Pregnancy Infections at the site of injection for the TPVB Allergy to dexamethasone; dexmedetomidine; ropivacaine Clinically significant cardiovascular, pulmonary, renal, or hepatic diseases

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-03-20 (Estimated); Primary Completion 2021-08-20 (Estimated); Study Completion 2021-08-30 (Estimated)

PRIMARY OUTCOMES:
the duration of analgesia | 48 hours after surgery
  time from completion of TPVB operation to VAS more than 3

SECONDARY OUTCOMES:
total sufentanil consumption | 48 hours after surgery
VAS | 1, 2, 4, 8, 12, 24, 36, and 48 hours after surgery
  VAS at rest and during coughing are evaluated by a blinded observer postoperatively
adverse effects | 48 hours after surgery

IPD SHARING:
Plan to Share IPD: Yes